CLINICAL TRIAL: NCT06125730
Title: A Single-Group Study to Evaluate the Effects of an Eyelash Serum on Improving Eyelash Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dime Beauty Co. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20362
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Eyelash Growth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DIME Beauty Eyelash Boost Serum (Experimental): Participants will use the eyelash serum twice daily in the morning and evening. The serum will be applied to the base of the top and bottom lashes.
  Interventions: Other: DIME Beauty Eyelash Boost Serum

INTERVENTIONS:
Other: DIME Beauty Eyelash Boost Serum — The test product contains Water, Glycerin, Amino Acids (Sodium PCA, Sodium Lactate, Arginine, Aspartic Acid, PCA, Glycine, Alanine, Serine, Valine, Proline, Threonine, Isoleucine, Histidine, Phenylalanine), Hyaluronic Acid, Panthenol, Aloe Leaf Extract, Niacinamide, Purslane, Chebulic Fruit Extract, Apple Fruit Extract, Tocopherol, Phenoxyethanol, Hexanediol, Ethylhexylglycerin, Biotinoyl Tripeptide-1, Myristoyl Pentapeptide-4.

SUMMARY:
This study will evaluate the efficacy of the DIME Beauty Eyelash Boost Serum in improving the growth of the eyelashes and their appearance in terms of length, fullness, and thickness. This study will last for 60 days. The study will be conducted as a single-arm trial in which all participants will use the test product. Participants will be required to undertake questionnaires at Baseline, Day 30, and Day 60, photos will be taken at Baseline, Day 30, and Day 60, and expert eyelash grading will take place at Baseline and Day 60.

ELIGIBILITY:
Inclusion Criteria:

Females aged 18-65. Wish to improve their eyelash growth. Wish to improve their eyelash length, thickness, and fullness. Have a smartphone or camera to take before-and-after selfies.

Exclusion Criteria:

Anyone not in good health. Anyone who has any chronic health conditions such as oncological or psychiatric disorders.

Anyone who has undergone any procedures that target the eyelashes in the past 3 months, or is planning to in the next 60 days. This includes eyelash lifts, tints, and extensions.

Anyone who has recently started using any product or taking any supplements that target eyelash growth, or who is planning to in the next 60 days.

Anyone who has any known serious allergic reactions that require the use of an Epi-Pen.

Anyone who is pregnant, breastfeeding, or wanting to become pregnant over the next three months.

Anyone who cannot/will not commit to the study protocol. Anyone with a history of substance abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Changes in eyelash growth as per expert grading. [Timeframe: Baseline to Day 60] | 60 days
  Before & after photos of the eyelashes will undergo grading by an eyelash expert.
Changes in participant-perceived eyelash growth. [Timeframe: Baseline to Day 60] | 60 days
  Measured via study-specific surveys. Surveys will be adapted from the validated Eyelash Satisfaction Questionnaire and designed on a 5-point Likert scale, with 5 representing the most favorable/best outcome (e.g., "Excellent") and 1 representing the least favorable/worst outcome (e.g., "Very poor").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided